CLINICAL TRIAL: NCT01918956
Title: A Prospective, Randomized, Open, Multi-centre Study to Assess Safety of PURETHAL Birch Given With a Rush Up-dosing Regimen to Patients With Allergic Rhinitis/Rhinoconjunctivitis
Brief Title: PURETHAL Birch RUSH Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: HAL Allergy (Industry)
Collaborators: Ergomed (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PB/0040
Record Dates: First submitted 2013-08-07; First posted 2013-08-08 (Estimated); Last update posted 2014-04-11 (Estimated); Status verified 2014-04

CONDITIONS: Allergic Rhinitis; Allergic Rhinoconjunctivitis
Keywords: immunotherapy; birch pollen; seasonal allergy; up-dosing
MeSH Terms: conditions — Rhinitis, Allergic; Rhinitis, Allergic, Seasonal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- conventional regimen of PURETHAL Birch (Active Comparator): Initial treatment:
  6 incremental weekly subcutaneous doses of 0.05, 0.1, 0.2, 0.3, 0.4 and 0.5 ml PURETHAL Birch, 20.000 AUM/ml (week 1, 2, 3, 4, 5, 6).
  Maintenance treatment:
  0.5 ml PURETHAL Birch, 20.000 AUM/ml, in intervals according to registered scheme (week 8, 10, 12).
  Interventions: Biological: PURETHAL Birch, 20.000 AUM/ml
- rush regimen of PURETHAL Birch (Experimental): Initial treatment:
  3 incremental weekly subcutaneous doses of 0.1, 0.3, and 0.5 ml PURETHAL Birch, 20.000 AUM/ml (week 1, 2, 3)
  Maintenance treatment:
  0.5 ml PURETHAL Birch, 20.000 AUM/ml, in 2-weekly intervals (week 5, 7, 9).
  Interventions: Biological: PURETHAL Birch, 20.000 AUM/ml

INTERVENTIONS:
Biological: PURETHAL Birch, 20.000 AUM/ml — comparison of different up-dosing regimes

SUMMARY:
This study investigates the safety of two up-dosing regimen. The safety of PURETHAL Birch will be evaluated in a rush regimen (maximum dose reached in 3 injections during 3 weeks) compared to the conventional regimen (maximum dose reached in 6 injections during 6 weeks).

The primary endpoint of the sudy is the comparison of the proportions of the patients who have successfully reached the maintenance dose between the two treatment regimes.

A similar previous study with PURETHAL Grasses has shown that the rush up-dosing scheme is as safe as the conventional up-dosing regime. Therefore it is expected that up-dosing with PURETHAL Birch according to the rush regimen is as safe as using the conventional regimen.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent.
* Age ≥12 years.
* Allergic rhinitis/rhinoconjunctivitis related to birch pollen with or without concomitant mild to moderate persistent asthma
* FEV1>70% for patients with a history of mild to moderate asthma, FEV1>70% or PEF>80% for patients without a history of asthma
* A positive SPT (mean wheal diameter ≥ 3mm compared to negative control and negative control should be negative) for birch pollen.
* Positive serum specific anti-birch IgE-test (>0.7 U/ml) within 1 year before randomization and/or a positive provocation test for birch pollen within 1 year before randomization.

Exclusion Criteria:

* Immunotherapy (SCIT or SLIT) with birch pollen allergens within the past 5 years
* Any specific immunotherapy (SCIT or SLIT) during the study period
* Severe immune disorders (including auto-immune diseases) and/or diseases requiring immunosuppressive drugs
* Active malignancies or any malignant disease within the past 5 years
* Severe uncontrolled diseases that could increase the risk for patients participating in the study
* Acute/active inflammation or infection of the target organs at the start of the study
* Secondary changes of the target organ
* Diseases with a contraindication for the use of adrenaline
* Use of systemic steroids within 4 weeks before start of the study and during the study
* Treatment with systemic and local β-blockers
* Vaccination within one week before start of therapy or during the initiation phase
* Anti-IgE therapy within the 6 months prior to inclusion and during the study
* Participation in a clinical study with a new investigational drug within the last 3 months or for a biological within the last 6 months prior to or during the study
* Pregnancy, lactation or inadequate contraceptive measures for women of child-bearing age
* Alcohol, drug or medication abuse within the past year
* Any clinically significant abnormal laboratory parameter at screening
* Lack or expected lack of cooperation or compliance
* Severe psychiatric, psychological, or neurological disorders
* Patients who are employees of the sponsor, institution or 1st grade relatives or partners of the investigator

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2013-09; Primary Completion 2014-02 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Proportion of patients successfully reaching the maintenance dose | 12 weeks

SECONDARY OUTCOMES:
Early and late local and systemic reactions | 30 minutes after IMP injection and 24 hours after injection
Immunological parameters (IgE, IgG) | 10 weeks rush regime, 13 weeks conventional regime

CONTACTS AND LOCATIONS:
Overall Officials: Piotr Buczyłko, Prof., Principal Investigator — NZOZ Centrum Alergologii
Locations (8):
- Poland (8):
  - NZOZ PROMEDICA Radlmacher i Wspólnicy Sp. J., Bialystok
  - NZOZ Alergia, Bielsko-Biala
  - NZOZ ClinicaVitae, Gdansk
  - Medica Pro Familia Sp.zo.o S.K.A, Katowice
  - ALERGO-MED.Specjalistyczna Przychodnia Lekarska Sp. z o.o., Tarnów
  - Specjalistyczne Centrum Medyczne CenterMed, Tarnów
  - NZOZ CUM PROXIMUM Sp. z o.o., Wroclaw
  - NZOZ Centrum Alergologii, Łódz